CLINICAL TRIAL: NCT02961075
Title: Impact of Local Anesthesia on Postbronchoscopy Fever: a Randomised Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: post2016taper
Record Dates: First submitted 2016-11-09; First posted 2016-11-10 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-11

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cricothyroid (Experimental): local surface anesthesia by Cricothyroid
  Interventions: Other: local surface anesthesia
- Laryngeal tube (Experimental): local surface anesthesia by Laryngeal tube
  Interventions: Other: local surface anesthesia; Device: Laryngeal tube

INTERVENTIONS:
Other: local surface anesthesia — Airway anesthesia for Bronchoscopy
Device: Laryngeal tube
  Arms: Laryngeal tube

SUMMARY:
Impact of Local Anesthesia on Postbronchoscopy Fever: a Randomised Controlled Study

DETAILED DESCRIPTION:
Fiberoptic bronchoscopy (FOB) is the essential procedures for diagnosis and treatment of respiratory diseases。 Fever following FOB has been frequently reported. Fever is usually caused by patient discomfort and delay recovery from illness, or even worse. The reported frequency of this complication ranges from 1 to 20%. According to previous reports, postbronchoscopy fever is associated with advanced age, the presence of abnormal bronchoscopic findings,documented endobronchial obstruction, bronchoscopic intervention for malignancy, BAL, bronchial brushing, endotoxin contamination during bronchoscopy, instillation of topical anesthetic through the bronchoscope, abnormal differential cell counts in the BAL fluid (BALF), bacterial growth in the BALF culture,and the severity of bleeding. At present, guidelines recommend sedation and analgesia combined with airway surface anesthesia for Fiberoptic bronchoscopy. laryngeal spray and cricothyroid anesthesia often used in clinical.Cricothyroid local anesthesia has a good effect, but it is an invasive operation, this is risk factors for fever after bronchoscopy.Therefore, to compare fever in the two kinds of airway anesthesia on Bronchoscopy . So as to provide the local anesthesia method with little influence on the patient.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III

Exclusion Criteria:

* use of immunosuppressive agents or corticosteroids
* body temperature 37.3°C during the 24 h prior to FOB,intubation or mechanical ventilation
* therapeutic bronchoscopy (foreign body removal, bronchial toilet, or stenting), discharge within 24 h of FOB
* surgical or diagnostic procedures within 24 h of FOB.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Fever | 48 hour
  Fever was defined as an axillary body temperature 37.3°C

CONTACTS AND LOCATIONS:
Overall Officials: Xiao z yang, MD,PhD, Study Director — 0866-17709873399
Locations (1):
- The Second Hospital of Dalian Medical University, Dalian, Liaoning, China